CLINICAL TRIAL: NCT01477632
Title: Single Dose, Three-way, Cross-over, Relative Bioavailability Study With 3 Oral Formulations for Hormone Replacement Therapy in Postmenopausal Women: 0.5 mg Estradiol + 0.1 mg Norethisterone Acetate, 0.5 mg Estradiol + 0.25 mg Norethisterone Acetate, and 1.0 mg Estradiol + 0.5 mg Norethisterone Acetate
Brief Title: Bioavailability of Three Oral Formulations for Hormone Replacement Therapy in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALD-1640; 2004-002457-32 (EudraCT Number)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Menopause; Healthy
MeSH Terms: interventions — Estradiol; Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: 0.5 mg estradiol / 0.1 mg norethisterone acetate (NETA)
- B (Experimental)
  Interventions: Drug: 0.5 mg estradiol / 0.25 mg norethisterone acetate (NETA)
- C (Active Comparator)
  Interventions: Drug: 1.0 mg estradiol / 0.5 mg norethisterone acetate (NETA)

INTERVENTIONS:
Drug: 0.5 mg estradiol / 0.1 mg norethisterone acetate (NETA) — A single oral dose of 2 tablets under fasting conditions
  Arms: A
Drug: 0.5 mg estradiol / 0.25 mg norethisterone acetate (NETA) — A single oral dose of 2 tablets under fasting conditions
  Arms: B
Drug: 1.0 mg estradiol / 0.5 mg norethisterone acetate (NETA) — A single oral dose of 1 tablet under fasting conditions
  Arms: C

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to determine the extent of bioavailability of two low dose estradiol/norethisterone acetate (NETA) preparations with a marketed estradiol/norethisterone acetate (NETA) preparation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Postmenopausal
* Caucasian race
* Smoking (up to 5 cig./per day) is allowed
* Good state of health: evidenced by medical history, physical examination including gynecological examination, results of laboratory examination

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Previous participation in this trial
* Previous estrogen and/or progestin hormone replacement therapy
* Known, suspected or history of breast cancer
* Systolic blood pressure (BP) at least 160 mm Hg and/or diastolic BP at least 100 mm Hg, currently treated or untreated
* Body Mass Index (BMI) above 35.0 kg/m^2

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC(0-∞))
Maximal concentration (Cmax)
Time to maximum (tmax)

SECONDARY OUTCOMES:
Area Under the Curve (AUC) from dosing up to last sample
Terminal half-life (t½)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neu-Ulm, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com